CLINICAL TRIAL: NCT00076973
Title: A Randomized, 2-Period, Multicenter, Dble-Blind, Parallel-Group Study Comparing Effects of 2 Doses of MK0476 and Placebo in the Tx of Respiratory Symptoms Associated w/ Respiratory Syncytial Virus-Induced Bronchiolitis in Children 3 to 24 Mths
Brief Title: An Investigational Drug Study to Treat Respiratory Symptoms Associated With Respiratory Syncytial Virus (RSV) Bronchiolitis (0476-272)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-272; Formerly 0112BRS; MK0476-272; 2004_098
Record Dates: First submitted 2004-02-06; First posted 2004-02-16 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Bronchiolitis
Keywords: RSV Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: montelukast sodium — Duration of Treatment: 6 months
  Other Names: MK0476
Drug: Comparator: placebo — Duration of Treatment: 6 months

SUMMARY:
The purpose of this study is to look at whether an investigational drug can treat the breathing symptoms of RSV bronchiolitis in children 3 to 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized or in an urgent/emergent-care setting at least 24 hours for a first or second episode of RSV-induced bronchiolitis. Approximately twenty percent of patients will be allowed in the study with a stay of less than 24 hours but need to meet a minimum predefined Respiratory Severity Score as required by the study.

Exclusion Criteria:

* Asthma or other wheezing disorder. The Primary Investigator will evaluate whether there are other reasons why a child may not participate.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1125 (Actual)
Dates: Start 2003-08; Primary Completion 2006-06 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Symptom-Free Days

SECONDARY OUTCOMES:
Percentage of Patients with Exacerbations and Percentage of Bronchiolitis-Free Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bisgaard H, Flores-Nunez A, Goh A, Azimi P, Halkas A, Malice MP, Marchal JL, Dass SB, Reiss TF, Knorr BA. Study of montelukast for the treatment of respiratory symptoms of post-respiratory syncytial virus bronchiolitis in children. Am J Respir Crit Care Med. 2008 Oct 15;178(8):854-60. doi: 10.1164/rccm.200706-910OC. Epub 2008 Jun 26. PMID 18583576